CLINICAL TRIAL: NCT03339310
Title: FIX-HF-5C2: Evaluation of the Safety and Efficacy of the 2-lead OPTIMIZER® Smart System in Subjects With Moderate-to-Severe Heart Failure With Ejection Fraction Between 25% and 45%
Brief Title: Evaluation of the Safety and Efficacy of the 2-lead OPTIMIZER® Smart System
Acronym: FIX-HF-5C2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Impulse Dynamics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP OPT2017-005; FIX-HF-5C2 (Other: Impulse Dynamics)
Record Dates: First submitted 2017-10-23; First posted 2017-11-13 (Actual); Last update posted 2020-01-14 (Actual); Status verified 2020-01

CONDITIONS: Heart Failure; Congestive Heart Failure; Chronic Heart Disease; CHF
Keywords: CCM Therapy; 2-Lead; FIX-HF-5C2; Optimizer
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: Optimizer Smart System
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Optimizer Smart System with 2-leads (Experimental): All eligible subjects will have the Optimizer Smart System implanted and receive cardiac contractility modulation therapy (CCM).
  Interventions: Device: Optimizer Smart System with 2-leads

INTERVENTIONS:
Device: Optimizer Smart System with 2-leads — The Optimizer Smart System with 2-leads delivers non-excitatory cardiac contractility modulating (CCM) electrical signals to the heart muscle. Implanted subjects receive five non-contiguous one-hour periods of CCM signals per day.
  Other Names: Optimizer Smart System

SUMMARY:
This is a multicenter, prospective, single-arm study of the Optimizer Smart System with 2-leads

DETAILED DESCRIPTION:
This is a multicenter, prospective, single-arm treatment only confirmatory study of the 2-lead configuration of the Optimizer Smart System.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are 18 years of age or older
* Subject is male or a non-pregnant female
* Subjects who have a baseline ejection fraction greater than or equal to 25% and less than or equal to 45% by echocardiography determined by the echocardiography core laboratory.
* Subjects who have been treated for heart failure for at least 90 days (including treatment with a β-blocker for at least 90 days unless the subject is intolerant) and are in New York Heart Association functional Class III and IV at the time of enrollment.
* Subjects receiving appropriate, stable medical therapy during the 30 days prior to enrollment for treatment of heart failure according to guideline recommendations. For patients with EF≤35%, this regimen shall consist of the appropriate doses of diuretics, ACE-inhibitor or angiotensin II receptor blocker and β-blocker. Angiotensin receptor -neprilysin inhibitor (ARNI) may be substituted for ACE inhibitors or ARBs and Ivabradine may also be considered in subjects with a heart rate >70bpm. Stable is defined as no more than a 100% increase or 50% decrease in dose.
* Subjects who, in the opinion of the Principal Investigator (based on the current guidelines for clinical practice), have a clinical indication for an implanted cardiac defibrillator (ICD, e.g., EF≤35%) and/or pacemaker, must have an existing device unless the patient refuses to undergo the implantation of such device for personal reasons.
* Subjects who are willing and able to return for all follow-up visits.

Exclusion Criteria:

* Subjects whose baseline peak VO2 is <9 or >20 ml O2/min/kg. The qualifying CPX test must be deemed adequate.
* Subjects who have a potentially correctible cause of heart failure, such as valvular heart disease or congenital heart disease.
* Subjects who have clinically significant angina pectoris, consisting of angina during daily life (i.e., Canadian Cardiovascular Society Angina score of II or more), an episode of unstable angina within 30 days before enrollment, or angina and/or ECG changes during exercise testing performed during baseline evaluation.
* Subjects hospitalized for heart failure requiring acute treatment with intravenous loop diuretics, IV inotropes or hemofiltration within 30 days before enrollment and baseline testing or subjects receiving any form of positive inotropic support within 30 days before enrollment, including continuous IV inotrope therapy.
* Subjects having a PR interval greater than 375ms.
* Subjects whose exercise tolerance is limited by a condition other than heart failure (e.g., angina, COPD, peripheral vascular disease, orthopedic or rheumatologic conditions) or who are unable to perform baseline stress testing.
* Subjects who are scheduled for a CABG or a PTCA procedure, or who have undergone a CABG procedure within 90 days or a PTCA procedure within 30 days of enrollment.
* Subjects who have a biventricular pacing system, an accepted indication for such a device, or a QRS width of 130ms or greater.
* Subjects who have had a myocardial infarction within 90 days of enrollment.
* Subjects who have mechanical tricuspid valve.
* Subjects who have a prior heart transplant.
* Subjects on dialysis.
* Subjects who are participating in another experimental protocol.
* Subjects who are unable to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-10-23 (Actual); Primary Completion 2019-10-30 (Actual); Study Completion 2019-10-30 (Actual)

PRIMARY OUTCOMES:
Change in exercise tolerance quantified by peak VO2 measured on cardiopulmonary exercise stress testing (CPX). | 24 weeks
  Device efficacy will be assessed as change in exercise tolerance quantified by peak VO2 measured on cardiopulmonary exercise stress testing (CPX). Subjects on device under FIX-HF-5C2 protocol will be compared to subjects on control under FIX-HF-5C protocol with respect to peak V02 mean change at 24-weeks from baseline.
Optimizer-device and -procedure related complication rate | 24 weeks
  Subjects experiencing an Optimizer device- or procedure-related complication through the 24-week study period, as determined by an independent events committee.

SECONDARY OUTCOMES:
Total CCM delivery comparing 2 and 3-lead device configurations | 24 weeks
  A comparison will be made between the Optimizer per-protocol groups in the FIX-HF-5C (3-lead) and FIX-HF-5C2 (2-lead) device configurations to show there is no difference between the amount of CCM therapy provided by the two device configurations. Total CCM delivery (effective hours delivered) will be evaluated at the end of 24 weeks following the Optimizer implantation.

CONTACTS AND LOCATIONS:
Overall Officials: David D. Gutterman, MD, Study Director — Medical College of Wisconsin
Locations (10):
- United States (9):
  - Chan Heart Rhythm Institute, Mesa, Arizona
  - Southwest Cardiology Associates, Mesa, Arizona
  - Cardiovascular Consultants, Phoenix, Arizona
  - Arizona Arrhythmia Consultants, Scottsdale, Arizona
  - Pima Heart Physicians, PC, Tucson, Arizona
  - Baptist Health Systems, Lexington, Illinois
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Dallas VA Hospital, Dallas, Texas
  - CHRISTUS Trinity Mother Frances, Tyler, Texas
- University Hospital gGmbH Bergmannsheil, Bochum, Germany

REFERENCES:
- [Derived] Wiegn P, Chan R, Jost C, Saville BR, Parise H, Prutchi D, Carson PE, Stagg A, Goldsmith RL, Burkhoff D. Safety, Performance, and Efficacy of Cardiac Contractility Modulation Delivered by the 2-Lead Optimizer Smart System: The FIX-HF-5C2 Study. Circ Heart Fail. 2020 Apr;13(4):e006512. doi: 10.1161/CIRCHEARTFAILURE.119.006512. Epub 2020 Apr 8. PMID 32264716